CLINICAL TRIAL: NCT03004092
Title: Novel Biomarkers for Invasive Aspergillosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The project with number S59863 has been completely transferred to S61979 - Hemoba
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S59863
Record Dates: First submitted 2016-12-21; First posted 2016-12-28 (Estimated); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Aspergillosis Invasive
Keywords: bis(methylthio)gliotoxin; lateral flow device; JF5; Galactomannan; Invasive aspergillosis
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Total cohort (Experimental)
  Interventions: Procedure: blood sample

INTERVENTIONS:
Procedure: blood sample — Twice weekly blood sample, and at every outpatient visit

SUMMARY:
Diagnosis of invasive aspergillosis remains difficult, and is often based on a combination of patient characteristics, radiological and microbiological findings. To data, galactomannan (GM) is the only well-validated biomarker available. However, GM still has its shortcomings. There is therefore a need for new, complementary biomarkers. In this study, two of those tests, bis(methylthio)gliotoxin (bmGT) and a lateral flow device, will be validated in a hematological population, and compare it to GM.

DETAILED DESCRIPTION:
Diagnosis of invasive aspergillosis is often difficult to achieve with certainty, as this requires direct evidence of invasive growth on histopathological examination. A probable diagnosis can be suspected based on both clinical and mycological evidence of the disease, in presence of a susceptible patient. The EORTC-MSG guidelines offer a widely accepted basis for this diagnosis. Under these guidelines, mycological evidence can consist of a positive culture of aspergillus spp, or of detection of galactomannan (GM) in a relevant body sample. GM is a part of the Aspergillus mould and can be detected using a commercially available immunoenzymatic sandwich microplate assay. However, like most biomarkers, galactomannan is far from a perfect biomarker. Several beta-lactam antibiotics are known to cause false positives, and anti-mould therapy has been reported to significantly lower the sensitivity[1]. Additional biomarkers that could circumvent these problems would therefore be beneficial.

A potential new target is gliotoxin (GT), a secondary metabolite of several fungi, the most clinically important of which is Aspergillus[2]. GT is released during invasive growth, and can therefore be used as a biomarker of invasive fungal disease by GT-producing fungi. However, GT is quickly removed by red blood cells from circulation, making it an unreliable marker[3]. A degradation product of GT, bis(methylthio)gliotoxin (bmGT), appears to be more stable as it is not taken up by red blood cells. Serum bmGT or bmGT in bronchoalveolar lavage (BAL) fluid has already been shown in small studies to be a potential marker of invasive aspergillosis, especially when used in combination with GM[3-5].

Recently, another highly specific test has become available, based on detection of an extracellular glycoprotein secreted during the growth of Aspergillus species, using a monoclonal antibody (JF5) in an immunochromatographic lateral-flow device (LFD)[6,7]. This test allows fast (<15 minutes) testing using a commercially available device.

In this study, both the LFD and bmGT will be characterized and validated in a hematological population, and compared to GM.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 16y at start of study
* One of the following diagnoses:
* De novo, refractory or relapsed AML/MDS receiving intensive chemotherapy
* De novo, refractory or relapsed ALL/T-lymphoblastic lymphoma receiving intensive chemotherapy
* Aplastic anemia requiring ATG therapy
* Any patient admitted for either autologous or allogeneic hematopoietic stem cell transplantation
* Written informed consent obtained from the patient

Exclusion Criteria:

* AML or ALL beyond the specified inclusion criteria
* Directed treatment for possible, probable, or proven invasive aspergillosis, at moment of screening, or with end of treatment < 6 weeks at screening, or no complete response according to EORTC/MSG criteria, or complete response achieved < 6 weeks at time of screening.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2017-01; Primary Completion 2019-12 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of serum bmGT | 2 weeks
  Determine the diagnostic accuracy (specificity, sensitivity predictive values, accuracy and other key diagnostic values) of serum bmGT in the diagnosis of invasive aspergillosis, using the revised EORTC criteria as gold standard.

SECONDARY OUTCOMES:
Diagnostic accuracy of a combination of serum bmGT and serum GM | 2 weeks
  Determine diagnostic accuracy of a combination of serum GM and serum bmGT in the diagnosis of invasive aspergillosis.
Prognostic value of serum bmGT | 6 weeks
  Determine prognostic value (therapy response / mortality) of initial serum bmGT levels.
Prognostic value of serum bmGT kinetics | 6 weeks
  Evaluate serum bmGT kinetics as surrogate marker of therapeutic response.
Renal and hepatic influence on bmGT | 2 weeks
  Evaluate the impact of renal and hepatic function on initial bmGT levels and bmGT kinetics.
Compare bmGT-HPTLC to bmGT-LC/MS | Same day
  Compare bmGT levels as measured by HPTLC to levels as measured by our own in-house developed chromatographic method.
Diagnostic accuracy of BAL bmGT | 2 weeks
  Determine diagnostic accuracy of bmGT in BAL in the diagnosis of invasive aspergillosis.
Diagnostic accuracy of LFD | 2 weeks
  Determine diagnostic accuracy of the lateral flow device (LFD) in BAL and serum in the diagnosis of invasive aspergillosis.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

REFERENCES:
- [Background] Pfeiffer CD, Fine JP, Safdar N. Diagnosis of invasive aspergillosis using a galactomannan assay: a meta-analysis. Clin Infect Dis. 2006 May 15;42(10):1417-27. doi: 10.1086/503427. Epub 2006 Apr 14. PMID 16619154
- [Background] Lewis RE, Wiederhold NP, Chi J, Han XY, Komanduri KV, Kontoyiannis DP, Prince RA. Detection of gliotoxin in experimental and human aspergillosis. Infect Immun. 2005 Jan;73(1):635-7. doi: 10.1128/IAI.73.1.635-637.2005. PMID 15618207
- [Background] Domingo MP, Colmenarejo C, Martinez-Lostao L, Mullbacher A, Jarne C, Revillo MJ, Delgado P, Roc L, Meis JF, Rezusta A, Pardo J, Galvez EM. Bis(methyl)gliotoxin proves to be a more stable and reliable marker for invasive aspergillosis than gliotoxin and suitable for use in diagnosis. Diagn Microbiol Infect Dis. 2012 May;73(1):57-64. doi: 10.1016/j.diagmicrobio.2012.01.012. Epub 2012 Apr 4. PMID 22480566
- [Background] Vidal-Garcia M, Domingo MP, De Rueda B, Roc L, Delgado MP, Revillo MJ, Pardo J, Galvez EM, Rezusta A. Clinical validity of bis(methylthio)gliotoxin for the diagnosis of invasive aspergillosis. Appl Microbiol Biotechnol. 2016 Mar;100(5):2327-34. doi: 10.1007/s00253-015-7209-6. Epub 2015 Dec 17. PMID 26678078
- [Background] Thornton CR. Development of an immunochromatographic lateral-flow device for rapid serodiagnosis of invasive aspergillosis. Clin Vaccine Immunol. 2008 Jul;15(7):1095-105. doi: 10.1128/CVI.00068-08. Epub 2008 May 7. PMID 18463222
- [Derived] Mercier T, Guldentops E, Lagrou K, Maertens J. Prospective Evaluation of the Turbidimetric beta-D-Glucan Assay and 2 Lateral Flow Assays on Serum in Invasive Aspergillosis. Clin Infect Dis. 2021 May 4;72(9):1577-1584. doi: 10.1093/cid/ciaa295. PMID 32188971